CLINICAL TRIAL: NCT07133542
Title: The 9-Box Performance Management Framework: Impacts on Body Weight Regulation and Exercise Behaviors in Graduate Students
Brief Title: A Waist Circumference and Body Fat Percentage Dual-Dimension Nine-Square Grid Model for Precision Obesity Management: A Randomized Controlled Trial in Overweight/Obese University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hainan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AQNU2024111
Record Dates: First submitted 2025-08-10; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Overweight and/or Obesity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Nine-Grid Matrix Group (Experimental): Tiered management via waist-risk/body-fat matrix. Participants receive bi-weekly health positioning and one of five precision strategies (e.g., high-intensity exercise + dietary control for Grid-I; low-intensity maintenance for Grid-IX). Real-time feedback via digital dashboard.
  Interventions: Behavioral: Dynamic Matrix Management for Weight Control (DMM-WC)
- Standard Aerobic Prescription Group (Placebo Comparator): Standardized progressive aerobic exercise at 40-90% heart rate reserve. Intensity/volume are personalized at baseline but remain static afterward. Adherence monitored using Huawei wearables (no dynamic adjustments or tiered feedback).
  Interventions: Behavioral: Standard Aerobic Prescription

INTERVENTIONS:
Behavioral: Dynamic Matrix Management for Weight Control (DMM-WC) — Precision weight management using a two-dimensional grid model. Participants undergo bi-weekly positioning on a waist risk-body fat matrix (9 grids), receiving tiered interventions (e.g., high-intensity exercise + dietary control for high-risk grids; maintenance plans for low-risk grids). Real-time progress feedback via visual spatial migration maps promotes adherence. Comparator group receives standardized aerobic prescription without dynamic adjustments.
  Arms: Dynamic Nine-Grid Matrix Group
Behavioral: Standard Aerobic Prescription — Personalized progressive aerobic exercise program. Participants receive baseline-adjusted intensity prescriptions (40-90% heart rate reserve), with adherence monitored via wearable devices. NO dynamic adjustments, tiered strategies, or visual feedback are provided throughout the 8-week intervention.
  Arms: Standard Aerobic Prescription Group

SUMMARY:
The goal of this randomized controlled trial is to test whether a dual-dimensional 9-grid matrix intervention improves body composition and exercise adherence compared to standard aerobic exercise in overweight/obese college students. The main questions it aims to answer are:

Does the 9-grid model optimize fat distribution (measured by waist-hip ratio) and sustain body fat reduction better than traditional exercise?

Does dynamic risk stratification in the 9-grid system enhance long-term exercise adherence?

How does spatial migration of participants within the grid (quantified by centroid index G) reflect intervention efficacy?

Researchers will compare the 9-grid management group (receiving dynamic positioning + 5-tier personalized strategies) to the control group (receiving standardized aerobic exercise) to see if the 9-grid model:

Reduces waist-hip ratio more effectively

Delays intervention plateau in body fat loss

Increases exercise adherence at 8 weeks

Participants will:

Undergo body measurements (weight, body mass index (BMI), body fat percentage, waist/hip circumference) at baseline, 4 weeks, and 8 weeks

Complete the Exercise Adherence Rating Scale (EARS) at 4 and 8 weeks

If in 9-grid group:

* Be classified into 1 of 9 grid zones every 2 weeks based on waist circumference risk + body fat status
* Receive zone-specific interventions (nutrition/exercise/behavioral guidance)

If in control group:

* Perform progressive aerobic exercise (40-90% heart rate reserve (HR) 3×/week
* Use heart rate monitors for intensity tracking

ELIGIBILITY:
Inclusion Criteria:

1. Age & Status:

   * Full-time university students aged 18-36 years
2. Overweight/Obesity Diagnosis (per Chinese criteria):

   * Males: Body Mass Index (BMI) ≥24 kg/m² AND waist circumference ≥85 cm
   * Females: Body Mass Index (BMI) ≥24 kg/m² AND waist circumference ≥80 cm
3. Exercise Capacity:

   * Able to safely perform moderate-intensity exercise (confirmed by Physical Activity Readiness Questionnaire [PAR-Q], all items "No")
4. Tech Compliance:

   * Own smartphone with proficiency in health apps (e.g., WeChat Sport)
5. Informed Consent:

   * Signed written consent with commitment to complete 12-week intervention

Exclusion Criteria:

1. Metabolic Diseases:

   * Diagnosed diabetes, thyroid dysfunction, or history of cardiovascular disease
2. Exercise Contraindications:

   * Orthopedic/neurological conditions limiting exercise
3. Confounding Medications:

   * Use of weight/metabolism-affecting drugs in past 3 months
4. Special Physiological Status:

   * Pregnancy or lactation
5. Conflicting Participation:

   * Concurrent enrollment in other weight-management trials

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-09 (Actual)

PRIMARY OUTCOMES:
Change in Waist-to-Hip Ratio (WHR) | Baseline, Week 4, Week 8
Body Mass Index (BMI) | Baseline, Week 8
Adherence to exercise | Week 4, Week 8
  Exercise adherence will be assessed using the standardized Exercise Adherence Rating Scale (EARS). This validated, self-reported questionnaire comprises 16 items. The first 6 items directly assess participants' behavioral adherence to the prescribed exercise regimen (e.g., session attendance, duration). The subsequent 10 items evaluate reasons for adherence or non-adherence, capturing key cognitive dimensions such as perceived barriers and motivation. All items are rated on a 5-point Likert scale ranging from "Completely Agree" (scored as 0) to "Completely Disagree" (scored as 4). Total scores are calculated such that higher scores indicate better exercise adherence.
Body Fat Percentage | Baseline, Week 4, Week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Hainan Normal University, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: Yes
1. Anthropometrics: Baseline/Week12 BMI, waist-hip ratio, body fat percentage
  2. Behavioral adherence: Weekly exercise adherence rating scalescores
  3. .Grid dynamics: Final nine-grid coordinate and migration distance
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 January 2030
Access Criteria: Academic researchers affiliated with accredited institutionsRegulatory bodies Peer reviewers for journal publication validationAccess Process:Step 1: Submit research proposal via OpenClinica PlatformStep 2: Institutional ethics approval documentation requiredStep 3: Data Use Agreement signing with corresponding authors
URL: https://www.openclinica.com

DOCUMENTS (1):
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT07133542/ICF_000.pdf